CLINICAL TRIAL: NCT02375347
Title: Effects of Adding Chickpeas to the American Diet on Fecal Microbiota Composition and Markers of Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: American Pulse Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 201400716
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Inflammation
Keywords: Gut Microbiota
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chickpea Enhanced Diet (Experimental): Fed an enhanced Chickpea diet over a short term period (Chickpea Enhanced Diet Short Term)
  Interventions: Other: Chickpea Enhanced Diet (Short term)

INTERVENTIONS:
Other: Chickpea Enhanced Diet (Short term) — Dry Roasted Chickpeas, 21.26 gram serving size bags, by mouth five times per week.
  Stool Samples collected at Day 1, Day 9, and Day 14.
  Other Names: Go'Bonzo's

SUMMARY:
This prospective study will assess the effects of adding legumes, especially chick peas, to the diet of healthy adults on the commensal bacteria from feces of human subjects and resulting self-reported GI symptoms as well as markers of immune function.

DETAILED DESCRIPTION:
Short-term active feeding study:

The investigators will provide various chickpea products to participants for a 14 day chickpea enhanced diet. Subjects will receive specific meal plan instructions for the consumption of 5 servings/week of chickpeas. Chickpea products will be sourced from commercial providers. While participants will be told to substitute chickpea products for other diet ingredients, the subjects will be free to choose what to substitute according to their preferences. Subjects will keep daily food records and will be told that chickpea consumption will be monitored in their fecal samples (qPCR). Fecal samples will be collected before the start (Day 1), during (Day 7-9) and at the end (Day 14) of the intervention using a stool collection kit (Sigma). Participants will complete our GI health questionnaire on a weekly basis to determine tolerance to increased chickpea intake. An open ended questionnaire will be administered after participants have completed the short-term study protocol to assess any issues with compliance to chickpea intake. All individuals that increased their chickpea intake from their usual diet by at least 3 servings/week will be included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Good Health
* No systemic antibiotics during the preceding two months
* No medication suppressing immune function
* Willingness to provide basic demographic as well as medical history data

Exclusion Criteria:

* Gastric Ulcers
* Inflammatory Bowel Disease (IBD) or Irritable Bowel Syndrome (IBS)
* Chronic constipation/diarrhea
* Body Mass Index (BMI) > 30
* Dietary restrictions that prevent legume intake
* Currently on any medication that can affect GI transit time
* Consumption of >3 servings/week of chickpeas or >6 servings/week of legumes BEFORE study begins

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Volker Mai, PhD, MPH, Principal Investigator — Associate Professor
Locations (1):
- Emerging Pathogens Institiute, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chickpea Enhanced Diet: Fed an enhanced Chickpea diet over a short term period (Chickpea Enhanced Diet Short Term)
  Chickpea Enhanced Diet (Short term): Dry Roasted Chickpeas, 21.26 gram serving size bags, by mouth five times per week.
  Stool Samples collected at Day 1, Day 9, and Day 14.
Period: Overall Study
Arm/Group | Chickpea Enhanced Diet
Started | 13
Completed | 12
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Chickpea Enhanced Diet
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Changes in Diversity of Gut Microbiota 16S rRNA Gene Sequences With Regard to Time.
Description: Compare the gut microbiota composition and overall diversity of individual subjects before and after the implementation of a controlled and observed diet of chickpeas and legume products, using 16S ribosomal RNA (rRNA) sequencing of fecal samples.
  The use of Operational Taxonomic Units (OTUs) are used to classify clusters of similar bacterial groups. OTUs are species or group of species often used when only DNA sequence data is available.
  This measure is the average amount of OTUs found for each time point.
Time Frame: Change in Baseline (Day 1, Day 7-9, and Day 14)
Measure: Mean (Standard Error); unit: Avg. Operational Taxonomic Units
Arm/Group | Chickpea Enhanced Diet
Number analyzed (Participants) | 12
Avg. Operational Taxonomic Units
  Baseline (Day 1) | 316.383 (78.249)
  Day 7-9 | 302.400 (89.735)
  Day 14 | 283.058 (85.620)

ADVERSE EVENTS:
Arm/Group | Chickpea Enhanced Diet
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chickpea Enhanced Diet (N=13)
Cracked Tooth (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No